CLINICAL TRIAL: NCT05879562
Title: Montreal Cognitive Assessment (MoCA) XpressO: Validation of a Digital Self-administered Cognitive Pre-screening Tool for the General Adult Population
Brief Title: Validation of a Digital Self-Administered Cognitive Screening Tool: MoCA-XpressO
Acronym: MoCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: MoCA Clinic and Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: MoCA Xpresso 01
Record Dates: First submitted 2023-05-16; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Cognitive Impairment; Cognitive Change; Cognitive Deficit; Assessment, Self
Keywords: Cognitive screening; Cognition; Cognitive impairment; Cognitive decline; Self-assessment
MeSH Terms: conditions — Cognitive Dysfunction; Cognition Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are blinded to which test is the one being validated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MoCA-Xpresso first (Experimental): Participants in the study will complete the MoCA-Xpresso test before the digital-MoCA classic test.
  Interventions: Diagnostic Test: MoCA-Xpresso
- MoCA-Xpresso second (Experimental): Participants in the study will complete the digital-MoCA classic test before the MoCA-Xpresso test.
  Interventions: Diagnostic Test: MoCA-Xpresso

INTERVENTIONS:
Diagnostic Test: MoCA-Xpresso — MoCA-Xpresso is a home-based, self-administered digital cognitive screening tool, based on a tablet device.

SUMMARY:
The investigators conducted a validation study for the Montreal Cognitive Assessment (MoCA)-XpressO compared to the digital-MoCA test (version 8.1) as the gold standard. Participants were recruited from the MoCA clinic and a family practice. Ethics approval was received, and all participants provided informed consent. A crossover study design was applied to the MoCA-XpressO and the digital-MoCA test; participants were randomized for the order of administration. The investigators only recruited participants who did not complete a MoCA test during the 3 months prior to the study. A logistic regression model was built, and the accuracy of the model was evaluated by the sensitivity, specificity, and area under the Receiver Operating Characteristic (ROC) curve.

DETAILED DESCRIPTION:
Introduction:

The MoCA XpressO is a self-administered medical digital cognitive screening test. This test can help individuals assess whether they should have concerns regarding their cognition and should bring these concerns up to their physician. The test can be administered in an empty office in the clinic, or in the comfort of the patient's home.

The MoCA Classic test was first published in 2005 by Nasreddine et al. (The Montreal Cognitive Assessment, MoCA: A Brief Screening Tool for Mild Cognitive Impairment. J Am Geriatr Soc, 2005, 53:695-9.) The MoCA Classic test (version 8.2) is a one-page 30-point test administered in 10 minutes. The test and administration instructions are freely accessible at www.mocatest.org. The test is available in over 55 languages and dialects. The MoCA Classic assesses several cognitive domains. The short-term memory recall task (5 points) involves two learning trials of five nouns and delayed recall after approximately 5 minutes. Visuospatial abilities are assessed using a clock-drawing task (3 points) and a three-dimensional cube copy (1 point). Multiple aspects of executive functions are assessed using an alternation task adapted from the trail-making B task (1 point), a phonemic fluency task (1 point), and a two-item verbal abstraction task (2 points). Attention, concentration and working memory are evaluated using a target detection task (1 point), a serial subtraction task (3 points), and a forward and backward digit sequence task (1 point each). Language is assessed using a three-item confrontation naming task with low- familiarity animals (3 points), a two-item syntactically complex sentence repetition task (2 points), and the aforementioned fluency task. Finally, orientation to time and place is evaluated (6 points).

Study objectives/purpose:

This study seeks to validate the MoCA XpressO self-administered digital test compared to the MoCA Classic test for adults aged 50+. The study's goal is to confirm its performance as a viable screening tool to flag concerns regarding cognition in this population.

Objectives and Hypotheses:

Primary Objective: establish validity by comparing the MoCA XpressO vs. the digital MoCA Classic test.

Validity Outcome 1: Correlation between the total score of MoCA XpressO and the total score of the digital MoCA Classic test.

Hypothesis 1: There will be a significant correlation between the total scores of the MoCA XpressO and MoCA Classic test.

Secondary Objective: explore the users' experience of the MoCA XpressO test through subjective feedback from the participant.

Outcome 2: subjective feedback about user experience for participant (Likert Scale) Hypothesis 2: user experience will be rated high (>=4) on a Likert scale 1-5.

Additional exploratory measures/data:

Demographic information (age, level of education etc.); diagnosis; previous MMSE or MoCA score if available; frequency of technological use

Study Sample: the target number of participants is 100. Participants will be recruited from the MoCA Memory Clinic and Institute and the Cornwall family practice clinic. Participants in this study will consist of adults age 50 and over, with no restrictions to sex, gender, or ethnicity. There will be an equal number of participants with normal cognition, mild cognitive impairment, and mild AD. They must speak English or French and have at least 6 years of formal schooling.

Study locations: 2 clinical sites will recruit potentially eligible participants. (1) MoCA Clinic and Institute, Greenfield Park, Québec, Canada; and (2) Family Medicine Practice, Cornwall, Ontario, Canada

Randomization:

The order of administration of the MoCA XpressO and the digital MoCA Classic test will be determined randomly so that each test will have similar chances of being first, or second. The same rater will be performing the MoCA Classic test in each clinic participating in the validation study.

Blinding: The participants are blinded to the screening test that is being studied. The researcher doing the analysis will be blinded to the order of randomization.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years and over
* All gender inclusive
* All sex inclusive
* Fluent in English or in French
* Minimum 6 years of formal education
* Minimum total score of 11/30 on MoCA test

Exclusion Criteria:

* Age younger than 50 years
* Less than 6 years of formal schooling
* Total score on MoCA test less than 11/30

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between the MoCA XpressO and the Digital MoCA | up to 30 minutes (for completion of all intervention included in the study)
  Correlation between the total score of MoCA XpressO and the total score of the Digital MoCA Classic

SECONDARY OUTCOMES:
Correlation between scores of sub-tests on MoCA-XpressO and the Digital MoCA | up to 30 minutes (for completion of all interventions in the study)
  Correlation between the scores of the sub-tests on MoCA XpressO and the scores of the sub-tests on the Digital MoCA Classic

CONTACTS AND LOCATIONS:
Overall Officials: Ziad Nasreddine, MD, Principal Investigator — MoCA Clinic and Institute, 4896 Taschereau Blvd bureau 230, Greenfield Park, Quebec J4V 2J2
Locations (1):
- MoCA Clinic and Institute, Greenfield Park, Quebec, Canada